CLINICAL TRIAL: NCT00353808
Title: An Open-Label Extension Trial Assessing The Safety And Tolerability Of [S,S]-Reboxetine In Patients With Postherpetic Neuralgia (PHN).
Brief Title: A Trial Assessing The Long Term Safety And Tolerability Of [S,S]-Reboxetine In Patients With Post-Shingles Pain.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been terminated early as the esreboxetine development program is being discontinued. There are no safety or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6061029
Record Dates: First submitted 2006-07-17; First posted 2006-07-19 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — O-methyl reboxetine

ARMS (1):
- s, s reboxetine (Experimental)
  Interventions: Drug: [S,S]-Reboxetine

INTERVENTIONS:
Drug: [S,S]-Reboxetine

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of [S,S]-Reboxetine in patients with chronic pain following shingles. This is the extension study of Protocol A6061026.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met the patient selection criteria for the preceding double-blind Protocol A6061026 and have completed the 16-week trial.
* Patients at screening must have a score of >/=40mm on the pain visual analogue scale.

Exclusion Criteria:

* Serious adverse event during the preceding double-blind Protocol A6061026 that was determined to be related to the trial medication by the Investigator.
* Patient treatment compliance was less than 80% in the preceding double-blind Protocol A6061026.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-07; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Vital signs
Physical examination
12-lead ECG
Hematology/Biochemistry
Adverse events

SECONDARY OUTCOMES:
Pain Visual Analogue Scale
Patient Global Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (56):
- United States (56):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Arcadia, California
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, Laguna Hills, California
  - Pfizer Investigational Site, Loma Linda, California
  - Pfizer Investigational Site, Redondo Beach, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Holly Hill, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Largo, Florida
  - Pfizer Investigational Site, Longwood, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Oak Brook, Illinois
  - Pfizer Investigational Site, Topeka, Kansas
  - Pfizer Investigational Site, Ruston, Louisiana
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Brockton, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Independence, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Nixa, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Amherst, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Orchard Park, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Canfield, Ohio
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Youngstown, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Tacoma, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061029&StudyName=A%20Trial%20Assessing%20The%20Long%20Term%20Safety%20And%20Tolerability%20Of%20%5BS%2CS%5D-Reboxetine%20In%20Patients%20With%20Post-Shingles%20Pain.%0D